CLINICAL TRIAL: NCT03849638
Title: Gait Analysis and Gait Training in Subjects 1 Year After Total Hip or Total Knee Replacement by Means
Brief Title: Gait Analysis and Gait Training in Patient With Total Hip or Total Knee Replacement
Acronym: WVPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Federica Bressi, MD, Campus Bio-Medico University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54/18 PAR ComEt CBM
Record Dates: First submitted 2019-02-15; First posted 2019-02-21 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip
Keywords: gait analysis; gait training; biofeedback

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gait training with real time biofeedback — Patients presenting asymmetry of the kinematic parameters of the step to the evaluation with sensorized treadmill, will undergo gait training program.
  The training program consists of 20 session (1 session/day) of gait training. Daily gait training will last 30 minutes as distributed:
  * 5 minutes of heating at a comfortable speed for the patient
  * Three 5-minute sessions of gait training with biofeedback interspersed with a break of 5 minutes each.

SUMMARY:
The main objective of the present study is the evaluation of the kinematic parameters of gait and distribution of the load, recorded thruogh a sensorized treadmill, on lower limbs in patients at 1 year from Total Hip Replacement or Total Knee Replacement.

The secondary objective is to evaluate the effects of gait training with biofeedback by means of a sensorized treadmill in patients with asymmetry of the kinematic parameters of the step and of distribution of the load on the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Examination ≥ 24
* 12 months after total hip or total knee replacement

Exclusion Criteria:

* impossibility to perform a walking test
* disabling cardiovascular and osteo-arthro-muscular problems that can impair walking tests
* central or peripheral neurological disorders that compromise the sensory-motor skills of the patient under examination and / or the degree of collaboration
* patients who have not signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait Speed | immediately after treatment
  meters/second
Step Length | immediately after treatment
  length in meters
Ground Contact Time | immediately after treatment
  Time in seconds
Hip Kinematics | immediately after treatment
  angles (degrees) of hip ROM
Knee Kinematics | immediately after treatment
  angles (degrees) of knee ROM
Ankle Kinematics | immediately after treatment
  angles (degrees) of ankle ROM
Lower limb loading | immediately after treatment
  load percentage distribution on lower limbs

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Department - Campus Bio-Medico University, Roma, RM, Italy